CLINICAL TRIAL: NCT05315219
Title: A Follow-up Study on the Long-term Treatment Effect and Quality of Life of Thyroid Cancer After Total Endoscopic Thyroidectomy Bilateral Areola Approach
Brief Title: A Follow-up Study on Total Endoscopic Thyroidectomy Bilateral Areola Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: 2021-0439
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Quality of Life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Thyroidectomy Bilateral Areola Approach (Experimental)
  Interventions: Procedure: Endoscopic Thyroidectomy Bilateral Areola Approach
- Open Thyroidectomy (No Intervention)

INTERVENTIONS:
Procedure: Endoscopic Thyroidectomy Bilateral Areola Approach — The endoscopic thyroidectomy achieves better cosmetic effects than open thyroidectomy, and is one of the most widely applied approach in China, meanwhile its safety and effectiveness has been broadly discussed since being introduced.
  Arms: Endoscopic Thyroidectomy Bilateral Areola Approach

SUMMARY:
Endoscopic thyroidectomy bilateral areola approach (ETBAA) is one of the most widely applied approach in China, meanwhile its safety and effectiveness has been broadly discussed since being introduced. However, these studies are generally with small sample size and short follow-up duration. The lack of long-term follow-up on oncological outcomes makes it inaccurate to evaluate the effectiveness of ETBAA versus OT. Thus, in this study, we evaluated long-term QoL and outcomes of patients with PTC underwent thyroidectomy via ETBAA versus OT.

ELIGIBILITY:
Inclusion Criteria:

* 1) Female patients under 55 years old; 2) no lateral cervical lymph node or distant metastasis were detected before the operation; 3) postoperative pathology confirmed the diagnosis of papillary thyroid carcinoma.

Exclusion Criteria:

* 1) Previous history of thyroid surgery; 2) lateral cervical lymph node dissection in the operation; 3) past or current history of underlying diseases including hyperthyroidism, hypertension, diabetes, coagulation dysfunction.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 295 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of life | 5 years
  measured by THYCA-QoL questionaire

IPD SHARING:
Plan to Share IPD: Undecided